CLINICAL TRIAL: NCT03213925
Title: Neoadjuvant Chemotherapy Followed by Radiotherapy Alone in Patients With Breast Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Instituto do Cancer do Estado de São Paulo (Other)
Responsible Party: Principal Investigator, Gustavo Nader Marta, Radiation Oncologist and Principal Investigator, Instituto do Cancer do Estado de São Paulo
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RT alone
Record Dates: First submitted 2017-07-08; First posted 2017-07-11 (Actual); Last update posted 2017-07-11 (Actual); Status verified 2017-07

CONDITIONS: Breast Cancer; Radiation Therapy
MeSH Terms: conditions — Breast Neoplasms | interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- RT (Experimental): After clinical response, breast magnetic resonance imaging (MRI) is performed and analyzed by two independent radiologists. Complete image response is defined by no enhanced tumor visible on any serial images.
  Radiation therapy to the breast with or without regional nodal area is performed within 12 weeks after completion of chemotherapy with conventional dose (25x200cGy). Additional boost of 16 Gy in the primary involved tumor region.
  Interventions: Radiation: Radiation therapy

INTERVENTIONS:
Radiation: Radiation therapy — Radiation therapy to the breast with or without regional nodal area is performed within 12 weeks after completion of chemotherapy with conventional dose (25x200cGy). Additional boost of 16 Gy in the primary involved tumor region.
  Techniques: 3D conformal radiation therapy or intensity modulated radiation therapy (IMRT).
  Standard systemic treatment for patients with hormonal positive receptor (hormone therapy for at least 5 years) and HER2 positive (trastuzumab for 1 year)

SUMMARY:
After neoadjuvant chemotherapy, patients normally receive either conservative breast surgery or mastectomy followed by radiation therapy. Some patients achieve a complete response after neoadjuvant chemotherapy. Considering that radiation therapy is an effective treatment for subclinical microscopic disease, the question arises whether breast surgery before radiation therapy can be avoided in the subgroup of patients with complete response after neoadjuvant chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Age 40 years or older
* Pathologically confirmed unicentric invasive breast cancer
* Clinical stage T1-3 / N0 or N2 / M0
* Clinical conditions to receive neoadjuvant chemotherapy

Exclusion Criteria:

* Prior diagnosis of cancer (exception: in situ cervical tumor and non-melanoma skin)
* Patient is known to be pregnant
* Prior history of radiation therapy in the thoracic region
* Impossibility to perform magnetic resonance imaging

Ages: 40 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Estimated)
Dates: Start 2017-06-01 (Actual); Primary Completion 2020-07-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Ipsilateral breast tumor recurrence (IBTR) | 5 years
  IBTR is defined from the date from complete response of neoadjuvant chemotherapy to the date of any ipsilateral locoregional recurrence or deth.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Radiology and Oncology of University of São Paulo - Radiation Oncology Unit, Instituto do Câncer do Estado de São Paulo (ICESP), Faculdade de Medicina da Universidade de São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No